CLINICAL TRIAL: NCT02992561
Title: Addressing Heightened Levels of Aggression in Traumatized Offenders With Psychotherapeutic Means: A Randomized Controlled Trial in Eastern DR Congo
Brief Title: Addressing Heightened Levels of Aggression in Traumatized Offenders With Psychotherapeutic Means
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Konstanz (Other)
Responsible Party: Principal Investigator, Anke Köbach, Postdoctoral Researcher, University of Konstanz
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FORNET1617
Record Dates: First submitted 2016-12-06; First posted 2016-12-14 (Estimated); Last update posted 2020-08-04 (Actual); Status verified 2020-07

CONDITIONS: Appetitive Aggression
Keywords: Aggression; Violence; Post-conflict reconstruction; Demobilization; Traumatized offenders
MeSH Terms: conditions — Aggression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Narrative Exposure Therapy (FORNET, adapted version) (Active Comparator): Version of Narrative Exposure Therapy for Forensic Offender Rehabilitation including one lifeline session and 5 exposure sessions as well as 6 group sessions adapted from behavioral-therapy approaches for addiction problems.
  Interventions: Behavioral: FORNET (adapted version)
- Waitlist control or treatment as usual (No Intervention): No intervention or non-specific measures of support on request

INTERVENTIONS:
Behavioral: FORNET (adapted version)
  Other Names: Narrative Exposure Therapy for Forensic Offender Rehabilitation (adapted version)
  Arms: Narrative Exposure Therapy (FORNET, adapted version)

SUMMARY:
Heightened levels of aggression are fuelling violent incidents at all levels, especially in post-war regions. Narrative Exposure Therapy for Forensic Offender Rehabilitation (FORNET) aims to address trauma symptoms along with reactive and instrumental/appetitive aggression to encounter the downward cycle of perpetration and enforce a sustainable (re-)integration into civil life. In the present study, the investigators provide an adapted version of FORNET to former combatants in the North Kivu, Eastern DR Congo. Structured baseline, 3 and 6 month follow up interviews will be administered to assess the main outcome measures recent violent acts and appetitive aggression.

DETAILED DESCRIPTION:
Participants will be recruited through local NGOs and eligible clients randomized to the treatment or waitlist control group, respectively. The treatment will be provided by supervised local counsellors after a 4-week training. At baseline, 3-month and 6-month follow up, sociodemographic data, trauma exposure, perpetrated violent acts, PTSD, recent aggression, functionality and drug dependency will be assessed. The interviews will be conducted by blind Congolese psychological interviewers after an intensive 3-weeks training and continuous supervision.

ELIGIBILITY:
Eligibility criteria

* Former participant of an armed group in DR Congo
* Involvement in violent attacks

Inclusion Criteria:

* PTSD diagnosis or AAS sum score of 22 or higher

Exclusion Criteria:

* Acute intoxification (alcohol or other drugs)
* Acute psychotic symptoms
* Sign of cerebro-organic diseases

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 402 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2019-03 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Appetitive aggression (sumscore; 0-60 indicating higher levels) | Change from baseline to 3-5 and 6-9 months post treatment
  Appetitive Aggression Scale (Weierstall & Ebert, 2011)
Current violent behavior (sumscore; 0-96 indicating more acts) | Change from baseline to 3-5 and 6-9 months post treatment
  A list of violent offenses perpetrated during the last 3 months (formerly used in Burundi; Crombach/Augsburger/Nandi)

SECONDARY OUTCOMES:
PSS-I: Posttraumatic Stress Disorder (sumscore, 0-80 indicating higher severity) | Change from baseline to 3-5 and 6-9 months post treatment
  PTSD Symptom Scale (Foa & Tolin, 2000)

OTHER OUTCOMES:
Social acknowledgement (0-45 indicating more social acknowledgment) | Change from baseline to 3-5 and 6-9 months post treatment
  Social Acknowledgement Questionnaire (Maerker & Mueller, 2004)
Depression (0-27 indicating higher severity) | Change from baseline to 3-5 and 6-9 months post treatment
  Patient Health Questionnaire - 9 (Kroenke & Spitzer, 2002)
Substance use problems | Change from baseline to 3-5 and 6-9 months post treatment
  Alcohol, Smoking and Substance Involvement Screening Test (Humeniuk et al., 2008)
Epigenetic changes | Change from baseline to 6-9 month post treatment
  Genome wide methylation patterns (to be explored)

CONTACTS AND LOCATIONS:
Overall Officials: Anke Köbach, PI, Principal Investigator — University of Konstanz
Locations (1):
- University of Konstanz, Konstanz, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Carleial S, Natt D, Unternahrer E, Elbert T, Robjant K, Wilker S, Vukojevic V, Kolassa IT, Zeller AC, Koebach A. DNA methylation changes following narrative exposure therapy in a randomized controlled trial with female former child soldiers. Sci Rep. 2021 Sep 16;11(1):18493. doi: 10.1038/s41598-021-98067-9. PMID 34531495
- [Derived] Koebach A, Carleial S, Elbert T, Schmitt S, Robjant K. Treating trauma and aggression with narrative exposure therapy in former child and adult soldiers: A randomized controlled trial in Eastern DR Congo. J Consult Clin Psychol. 2021 Mar;89(3):143-155. doi: 10.1037/ccp0000632. PMID 33829803
- [Derived] Robjant K, Koebach A, Schmitt S, Chibashimba A, Carleial S, Elbert T. The treatment of posttraumatic stress symptoms and aggression in female former child soldiers using adapted Narrative Exposure therapy - a RCT in Eastern Democratic Republic of Congo. Behav Res Ther. 2019 Dec;123:103482. doi: 10.1016/j.brat.2019.103482. Epub 2019 Sep 27. PMID 31639529
- See also: Results for the group of female former child soldiers — https://doi.org/10.1016/j.brat.2019.103482